CLINICAL TRIAL: NCT00743184
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Trial of the Safety and Efficacy of Ozarelix, in Patients With Lower Urinary Tract Symptoms (LUTS) Due to Benign Prostatic Hyperplasia (BPH)
Brief Title: Trial of the Safety and Efficacy of Ozarelix in Participants With Benign Prostatic Hyperplasia (BPH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPI-153-08-1
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Benign Prostatic Hyperplasia (BPH); Lower Urinary Tract Symptoms (LUTS)
Keywords: BPH; LUTS; Lower urinary tract symptoms (LUTS)
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — ozarelix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo + Placebo (Placebo Comparator): Participants will receive Placebo + Placebo on Days 0 and 14 of each 6-month course.
  Interventions: Drug: Placebo
- 15 mg Ozarelix + 15 mg Ozarelix (Experimental): Participants will receive 15 mg Ozarelix + 15 mg Ozarelix on Days 0 and 14 of each 6-month course.
  Interventions: Drug: ozarelix
- 30 mg Ozarelix + 15 mg Ozarelix (Experimental): Participants will receive 30 mg Ozarelix + 15 mg Ozarelix on Days 0 and 14 of each 6-month course.
  Interventions: Drug: ozarelix

INTERVENTIONS:
Drug: ozarelix — One single-dose vial contains 16.5 mg of ozarelix. The drug is reconstituted with 1.3 mL of diluent.
  Arms: 15 mg Ozarelix + 15 mg Ozarelix; 30 mg Ozarelix + 15 mg Ozarelix
Drug: Placebo — Identical placebo is also provided and reconstituted using diluent containing 0.1% saline solution.
  Arms: Placebo + Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled study to evaluate the efficacy of ozarelix compared to placebo in the treatment of lower urinary tract symptoms (LUTS) secondary to benign prostatic hyperplasia (BPH) in men as assessed by the International Prostate Symptom Score (IPSS) at Week 14.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled study.

Participants who meet the entry IPSS inclusion criteria at Week 0 will be randomized and enroll in the double-blind treatment period. Participants will be randomized to one of three treatment arms and will receive two 6-month courses of study drug administered on Days 0 and 14 of each 6-month course. Treatment arms include: ozarelix 30mg + 15mg, ozarelix 15mg + 15mg or placebo + placebo. Safety and efficacy assessments will be performed at defined intervals throughout the study. At Week 52 all participants on study will be eligible to receive ozarelix for two additional courses in the open-label treatment period.

ELIGIBILITY:
Inclusion Criteria (All must be answered yes):

1. Has the participant given written informed consent?
2. Is the participant at least 50 years old?
3. Is the participant diagnosed with BPH and has he had clinical signs and symptoms of BPH for ≥ 6 months?
4. Does the participant have an IPSS ≥ 13?
5. Does the participant have a peak urinary flow rate (Qmax) of 4-15 mL/sec (utilizing the 2-second rule) established on a voided volume of at least 125 mL?
6. Does the participant have an IPSS Quality of life (QoL) score of ≥ 3?
7. Does the participant have a PSA > 0.8 ng/mL?
8. For participant with a PSA between 4 and 10 ng/mL or suspicion of prostate cancer, has the patient had a diagnostic evaluation (e.g., biopsy, PSA, velocity, etc.) that reasonably excludes the diagnosis of prostate cancer?
9. Is the participant willing to agree not to use any other approved or experimental pharmacologic BPH treatments including but not limited to alpha blockers, 5-alpha reductase inhibitors, anti-cholinergic preparations or herbal preparations at any time during the study?
10. Is the participant willing to restrict use of Phosphodiesterase 5 (PDE 5) inhibitors exclusively to the use of Viagra, one dose per week only and with no dosing in the 5 days immediately preceding scheduled study visit?
11. Is the patient willing and able to abide by the protocol?
12. Does the participant have an IPSS ≥ 13?
13. Does the participant have an IPSS QoL score of ≥ 3?
14. Does the participant have a post-void residual ≤ 350cc?

Exclusion Criteria (all must be answered No):

1. Does the participant have a history of prostate cancer or a serum prostate specific antigen (PSA) >10 nanogram per milliliter (ng/mL)?
2. Has the participant had prior prostate or bladder surgery, pelvic surgery (excluding hernia repair), pelvic radiation or lower urinary tract malignancy?
3. Does the participant have a prevoid total bladder volume assessed by ultrasound > 550 mL?
4. Does the participant have a post void residual urine volume ≥ 350 mL by ultrasound?
5. Has the participant taken or is the patient currently taking any of the following:

   1. Estrogens, phytoestrogens, androgens, antiandrogens or luteinizing hormone-releasing hormone (LHRH) agonists within the past 4 months (e.g. testosterone gel [Androgel ®1%, Testim ® 1%], testosterone buccal [Striant®], oxymetholone [Anadrol®-50], oxandrolone [Oxandrin®], esterified estrogen and methyltestosterone [Estratest®]), bicalutamide [Casodex®], nilutamide [Nilandron®], flutamide [Eulexin®], leuprolide acetate [Lupron®, Eligard®, Viadur®], goserelin acetate [Zoladex®] or,
   2. 5 α-reductase inhibitors within the past 4 months (e.g. finasteride[Proscar®, Propecia®], dutasteride [Avodart®]) or,
   3. Alpha blockers or anti-cholinergic preparations within the past 6 weeks (e.g. doxazosin [Cardura®], terazosin [Hytrin®], tamsulosin [Flomax®], alfuzosin [Uroxatrol®], oxybutynin [Ditropan®], tolterodine [Detrol-LA®], amitriptyline [Elavil®, Limbitrol®]) or,
   4. Class 1A (e.g. quinidine, procainamide, disopyramide) or Class III Anti-arrhythmic (e.g.sotalol [Betapace®], amiodarone [Cordarone®])
6. Does the participant have or has the patient ever had a diagnosis of acute or chronic prostatitis or chronic pelvic pain syndrome?
7. Has the participant had a urinary tract infection or instrumentation (e.g catheterization, cystoscopy, prostate biopsy) within the past 4 weeks?
8. Does the participant have a history of urethral stricture, bladder stones, obstructing median lobe or neurogenic bladder dysfunction?
9. Does the participant have microscopic hematuria greater than trace by dipstick urine at Visit 1?
10. Did the participant have a positive drug screening result?
11. Does the participant have a history of urinary retention?
12. Does the participant have any serious medical condition (e.g., Congestive heart failure [CHF], poorly controlled diabetes (Hemoglobin A1C [HgbA1c] > 9), psychiatric disorder, drug or alcohol abuse) that might interfere with his ability to comply with or complete the protocol?
13. Is the participants corrected QT interval (QTc) interval on the screening electrocardiogram (ECG) > 450ms, or does he have a family history of long QT syndrome?
14. Does the participant anticipate or plan to have an elective surgery or surgical procedure requiring general, spinal or epidural anesthesia during the course of the double-blind treatment portion of the study(within the next 12 months)?
15. Has the participant ever received ozarelix, cetrorelix, teverelix or degarelix?
16. Has the participant participated in any other study of an investigational drug or treatment for the signs and symptoms LUTS or BPH in the past 12 months?
17. Has the participant participated in any other clinical research study or study of an investigational drug in the past 90 days?

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-12-04 (Actual); Primary Completion 2010-01-20 (Actual); Study Completion 2010-01-20 (Actual)

PRIMARY OUTCOMES:
Change From Baseline International Prostate Symptom Score (IPSS) Score at Week 14 | Week 14
  IPSS is a validated self-administered index for grading benign prostatic hyperplasia (BPH)-related signs and symptoms. It consists of a set of seven questions. A total score of 1-7 indicates mild disease, 8-19 moderate disease and 20-35 severe disease.

SECONDARY OUTCOMES:
Change From Baseline IPSS (Including Sub-scores) at Week 52 | Week 52
  The International Prostate Symptom Score (IPSS) consists of 7 questions concerning urinary symptoms and 1 question concerning quality of life (QoL) with total score and subscores (voiding, storage and QoL). 1) Voiding- The subscale voiding score is the sum of the responses to 4 voiding symptoms questions (incomplete emptying, intermittency, weak stream, and straining). 2) Storage- The subscale storage score is the sum of the responses to 3 storage symptoms questions (frequency, urgency, and nocturia). Voiding and Storage: the lowest and highest possible scores range from 0 to 15 (mildly symptomatic to severely symptomatic). Voiding and Storage: each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. And 3) QoL assessment was a single question asking the participant how he would feel about tolerating his current level of symptoms for the rest of his life. The lowest and highest possible score ranges from 0 to 6 (very pleased to terrible).
Change From Baseline Benign Prostatic Hyperplasia Impact Index (BPHII) Score at Week 14 and Week 52 | Weeks 14 and 52
  BPH Impact Index (BII) is used to assess the impact of BPH on various aspects of health. This 4 question self administered index uses a scoring range from 0 (best) to 13 (worst).
Lower Urinary Tract Symptoms (LUTS) Global Assessment Question (LUTS-GAQ) Response at Week 52 | Week 52
  The self administered LUTS GAQ is a "yes" or "no" response to a question asking whether overall improvement in LUTS will be observed during the treatment period.
Change From Baseline Maximum Urine Flow (Qmax) at Week 14 and Week 52 | Week 14 and Week 52
  Qmax was measured by free flow uroflowmetry. Qmax is defined as the peak urine flow rate (measured in milliliter (mL)/second using a standard calibrated flowmeter). For a Qmax to be considered valid, the voided volume had to be at least 125 mL. The uroflowmeter is to be calibrated weekly.
Change From Baseline International Index of Erectile Function-15 (IIEF-EF) Score at Week 14 and Week 52 | Week 14 and Week 52
  IIEF-EF is defined as the sum of the scores for Questions 1-5 and 15 of the IIEF questionnaire. This recall instrument is self-administered by the participant. Individual questions are graded from 1 to 5 with a maximum total score of 30. Lower IIEFEF scores represent diminished erectile function. Men with a score of ≥ 26 are interpreted as having normal erectile function.
Change From Baseline International Prostate Symptom Score - Quality of Life (IPSS-QOL) at Week 14 and Week 52 | Week 14 and Week 52
  IPSS QOL is a disease-specific quality of life question, referred to as IPSS Question 8. Participants with an IPSS QOL of <3 at screening will be excluded from this study. The rating is as follows: 0=delighted, 1=pleased, 2=mostly satisfied, 3=mixed, 4=mostly dissatisfied, 5=unhappy, 6=terrible.
Number of Participants With Treatment-Emergent Adverse Events | Up to 104 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- California Professional Research, Newport Beach, California, United States